CLINICAL TRIAL: NCT06513481
Title: A Study of Enhancing Drug Prophylaxis of Venous Thromboembolism in Chinese Colorectal Cancer Surgery: a Multicenter, Prospective, Observational Cohort Study
Brief Title: A Study of Enhancing Drug Prophylaxis of Venous Thromboembolism in Chinese Colorectal Cancer Surgery
Acronym: E-DISTANCE
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Zhi-chun Gu, associate professor of pharmacy, RenJi Hospital
Other Study IDs: LY-007-B-AMD-01
Record Dates: First submitted 2024-07-17; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and Colorectal cancer tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early initiation of drug prophylaxis (within 24 hours after surgery): Patients who underwent surgery received prophylactic administration of low molecular weight heparin (nardraparin calcium injection) at a time point of 24 hours after surgery，this group carries out early initiation of drug prophylaxis (within 24 hours after surgery)
  Interventions: Drug: Nardraparin calcium injection
- Late initiation of drug prophylaxis (24 hours after surgery): Patients who underwent surgery received prophylactic administration of low molecular weight heparin (nardraparin calcium injection) at a time point of 24 hours after surgery，this group carries out late initiation of drug prophylaxis ( 24 hours after surgery)
  Interventions: Drug: Nardraparin calcium injection

INTERVENTIONS:
Drug: Nardraparin calcium injection — The dose of nardraparin calcium injection is 100AxaIU/kg, adjusted according to the patient's body weight, and is injected subcutaneously once a day
  Groups: Early initiation of drug prophylaxis (within 24 hours after surgery)
Drug: Nardraparin calcium injection — The dose of nardraparin calcium injection is 100AxaIU/kg, adjusted according to the patient's body weight, and is injected subcutaneously once a day
  Groups: Late initiation of drug prophylaxis (24 hours after surgery)

SUMMARY:
This project intends to conduct a multicenter, prospective, observational cohort study, aiming to explore the impact of the timing of pharmacological thromboprophylaxis initiation on postoperative bleeding risk and the effectiveness of venous thromboembolism (VTE) prevention in Chinese patients after colorectal cancer (CRC) surgery. The research outcomes of this project could provide valuable insights for optimizing the prevention and management of VTE after CRC surgery.

ELIGIBILITY:
Inclusion Criteria:

- 1.Age > 18 years old; 2.The patient was diagnosed with colorectal cancer, and the cTMN stage was cT1-2, N0 or cT3, N0 or any cT, N1-2； 3.The patient was diagnosed with colorectal cancer and was able to receive radical surgery (laparoscopic or open surgery). The expected operation time was >45 minutes, and the expected postoperative survival time was >6 months.

4.The patient or guardian agrees to the study plan and signs the informed consent.

Exclusion Criteria:

* 1.Renal insufficiency (CrCl<30 mL/min) or hepatic insufficiency (ALT> 3 times the upper limit of normal); 2.The patient was diagnosed with colorectal cancer with a cTMN stage of cT4 and/or local unresectable lesions. Unresectable local recurrent lesions included: (1) extensive lateral pelvic wall invasion, (2) external iliac vascular involvement, (3) tumor invasion into the great sciatic notch, sciatic nerve invasion, and (4) invasion of the second sacrum level and above.

  3.Known allergy to low molecular weight heparin (LWMH), narcotic drugs or radiocontrast agents; 4.The presence of systemic hemorrhagic disease or bleeding tendency, such as active peptic ulcer, uncontrolled hypertension, cerebral thrombosis, cerebral hemorrhage or neurosurgical history within 6 months; 5.Known brain metastases, endocarditis, or history of heparin-induced thrombocytopenia; 6.VTE occurred within 3 months before surgery; 7.Use heparin or oral anticoagulant therapy within 5 days before surgery; 8.Women who are pregnant or breastfeeding; 9.Any situation in which the investigator determines that the subject is not suitable for anticoagulant therapy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients were diagnosed with colorectal cancer and underwent radical surgery (laparoscopic or open surgery) with an estimated operation time of >45 minutes. Patients with expected survival >6 months after surgery.
Sampling Method: Probability Sample
Enrollment: 914 (Estimated)
Dates: Start 2024-07-16 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
VTE events within 28 days after surgery | 7 and 28 days after surgery
  Patients were followed up for VTE events, including deep vein thrombosis (DVT) and pulmonary thromboembolism (PE), within 28 days after surgery. Diagnosis of DVT: The lower limb is examined based on clinical symptoms (swelling and pain in the lower limb, tenderness in the back of the lower limb and/or in the inner thigh) and/or by color ultrasound or venography. The diagnosis of PE is based on clinical findings (dyspnea and shortness of breath), laboratory tests (plasma D-dimer), and CT pulmonary angiography (CTPA). Vte events were evaluated at 7 and 28 days after surgery. If a patient develops a VTE event, the patient is treated with VTE and assessed for thrombotic progression by ultrasound in both lower limb veins after 2 weeks.

SECONDARY OUTCOMES:
Any bleeding event within 28 days after surgery | 1，3，7 and 28 days after surgery
  Patients were followed up for any bleeding events within 28 days after surgery, including major and minor bleeding events. According to the International Society of Thrombosis and Hemostasis Standards (ISTH standards). All patients were followed up at 1, 7, and 28 days after surgery through inpatient or outpatient follow-up and bleeding investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Chun Gu, Principal Investigator — Department of Pharmacy, Renji Hospital, School of Medicine, Shanghai Jiao Tong University

IPD SHARING:
Plan to Share IPD: Undecided